CLINICAL TRIAL: NCT02318706
Title: An Asian, Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled 14-Week Study of DS-5565 in Patients With Diabetic Peripheral Neuropathic Pain Followed by a 52-Week Open-label Extension
Brief Title: DS-5565 Phase III Study for Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry); Quintiles, Inc. (Industry); Quintiles Malaysia Sdn Bhd (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS5565-A-J303
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — mirogabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo (Placebo Comparator): placebo group (14 weeks)
  Interventions: Drug: placebo
- DS-5565 15mg (Experimental): DS-5565 15 mg, oral administration, Treatment period; 2-weeks titration and 12-weeks fixed dose
  Interventions: Drug: DS-5565
- DS-5565 20 mg group (Experimental): DS-5565 20 mg, oral administration, Treatment period; 1-week titration and 13-weeks fixed dose
  Interventions: Drug: DS-5565
- DS-5565 30 mg group (Experimental): DS-5565 30 mg, oral administration, Treatment period; 2-weeks titration and 12-weeks fixed dose
  Interventions: Drug: DS-5565

INTERVENTIONS:
Drug: DS-5565
  Other Names: mirogabalin
  Arms: DS-5565 15mg; DS-5565 20 mg group; DS-5565 30 mg group
Drug: placebo
  Arms: placebo

SUMMARY:
Investigate the efficacy and safety of DS-5565 in subjects with Diabetic Peripheral Neuropathic Pain (DPNP) in comparison to placebo

DETAILED DESCRIPTION:
[Double Blind Phase] The primary objective is to compare change in the Average Daily Pain Score(ADPS) from baseline to Week 14 in Asian subjects with DPNP receiving DS-5565 versus placebo.

[Open Extension Phase] The objective is to assess the long-term safety and efficacy of DS-5565 in subjects with DPNP.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus at screening
* Painful distal symmetric polyneuropathy
* At screening, a pain scale of ≥ 40 mm

Exclusion Criteria:

* HbA1c (National Glycohemoglobin Standardization Program) > 10.0%

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Saiki Central Hospital, Ōita, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Kato J, Baba M, Kuroha M, Kakehi Y, Murayama E, Wasaki Y, Ohwada S. Safety and Efficacy of Mirogabalin for Peripheral Neuropathic Pain: Pooled Analysis of Two Pivotal Phase III Studies. Clin Ther. 2021 May;43(5):822-835.e16. doi: 10.1016/j.clinthera.2021.03.015. Epub 2021 May 29. PMID 34059327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 854 participants who met all inclusion and no exclusion criteria were enrolled; 834 were randomized to treatment in the double-blind phase. Twenty participants were excluded by the sponsor due to a serious Good Clinical Practice violation (inform consent form-related). A total of 214 participants enrolled in the open-label extension.
Pre-assignment Details: Participants were randomized to DS-5565 (15, 20, or 30 mg) or placebo in the double-blind (DB) phase and open-label DS-5565 in the long-term (LT) phase. Patients who complete the DB phase may not enroll in the LT phase. DB phase determine significant difference vs placebo (~750 target cases). LT phase confirm long-term safety (~180 target cases).
Groups:
- Placebo: Participants who received an oral dose of placebo twice daily (BID) for 14 weeks.
- DS-5565 15mg QD: Participants who received an oral dose of DS-5565 15 mg every day (QD).
  During the titration period, DS-5565 was administered orally at a daily dose of 5 mg (5 mg QD) during the first week and followed by 10 mg (10 mg QD) during the second week.
  During the fixed-dose period, a daily dose of 15 mg (15 mg QD) was administered orally for 12 weeks.
- DS-5565 20 mg (10 mg BID): Participants who received an oral dose of DS-5565 20 mg (10 mg BID).
  During the titration period, DS-5565 was administered orally at a daily dose of 10 mg (5 mg BID) for 1 week.
  During the fixed-dose period, a daily dose of 20 mg (10 mg BID) was administered orally for 13 weeks.
- DS-5565 30 mg (15 mg BID): Participants who received an oral dose of DS-5565 30 mg (15 mg BID).
  During the titration period, DS-5565 was administered orally at a daily dose of 10 mg (5 mg BID) for the first week followed by 20 mg (10 mg BID) during the second week.
  During the fixed-dose period, a daily dose of 30 mg (15 mg BID) was administered orally for 12 weeks.
- DS-5565 Open-label Extension: Participants who received an oral dose of DS-5565 5 mg BID for the first 2 weeks and 10 mg BID for the second 2 weeks (i.e., Week 3 and 4). At Week 5, the dosage was escalated to 15 mg BID if there were no concerns in safety. For the subsequent visits, the dosage may have changed to either 10 mg BID or 15 mg BID depending on safety findings.
Period: Double-blind Phase
Arm/Group | Placebo | DS-5565 15mg QD | DS-5565 20 mg (10 mg BID) | DS-5565 30 mg (15 mg BID) | DS-5565 Open-label Extension
Started | 334 | 166 | 168 | 166 | 0
Completed | 309 | 154 | 150 | 142 | 0
Not Completed | 25 | 12 | 18 | 24 | 0
Not completed — Adverse Event | 7 | 4 | 3 | 10 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 2 | 4 | 3 | 0
Not completed — Withdrawal by Subject | 9 | 5 | 7 | 10 | 0
Not completed — Other | 4 | 1 | 2 | 1 | 0
Not completed — Death | 0 | 0 | 2 | 0 | 0
Period: Open-label Extension Phase
Arm/Group | Placebo | DS-5565 15mg QD | DS-5565 20 mg (10 mg BID) | DS-5565 30 mg (15 mg BID) | DS-5565 Open-label Extension
Started | 0 | 0 | 0 | 0 | 214 (A portion of participants who completed the double-blind phase enrolled in the open-label extension.)
Completed | 0 | 0 | 0 | 0 | 172
Not Completed | 0 | 0 | 0 | 0 | 42
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 21
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 19

BASELINE CHARACTERISTICS:
Groups:
- DS-5565 15mg QD: Participants who received an oral dose of DS-5565 15 mg QD.
  During the titration period, DS-5565 was administered orally at a daily dose of 5 mg (5 mg QD) during the first week and followed by 10 mg (10 mg QD) during the second week.
  During the fixed-dose period, a daily dose of 15 mg (15 mg QD) was administered orally for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | DS-5565 15mg QD | DS-5565 20 mg (10 mg BID) | DS-5565 30 mg (15 mg BID) | Total
Number analyzed (Participants) | 334 | 166 | 168 | 166 | 834
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 198 | 99 | 102 | 98 | 497
  >=65 years | 136 | 67 | 66 | 68 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (10.5) | 61.9 (8.4) | 61.2 (10.1) | 61.8 (9.4) | 61.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 53 | 47 | 36 | 229
  Male | 241 | 113 | 121 | 130 | 605
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 334 | 166 | 168 | 166 | 834
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 334 | 166 | 168 | 166 | 834
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in the Average Daily Pain Score (ADPS) From Baseline to Week 14 Following Administration of DS-5565 in Participants With Diabetic Peripheral Neuropathic Pain
Description: Each participant recorded a pain score in the electronic patient diary once daily from the day after the screening visit (Visit 1) to the end of treatment/early termination visit (Visit 10). Prior to taking the study drug each morning, the participant selected the number that best described his or her pain over the past 24 hours on a scale of 0 (no pain) to 10 (worst possible pain). Higher ADPS scores indicated worse outcome. ADPS was the weekly average pain score based on the pain scores from the electronic patient diaries (Pain diary).
  In this outcome, the change from baseline in ADPS is being reported with negative values representing improvements in average daily pain. The larger the negative value (ie. improvement), the greater the improvement in average daily pain.
Time Frame: Baseline to Week 14 (post-dose 1 [15 mg QD] and post-dose 2 [20 mg and 30 mg])
Population: ADPS was assessed in the Modified-Intent-to-Treat Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | DS-5565 15mg QD | DS-5565 20 mg (10 mg BID) | DS-5565 30 mg (15 mg BID)
Number analyzed (Participants) | 330 | 164 | 165 | 165
units on a scale
  Week 1 | -0.26 (0.79) | -0.39 (0.67) | -0.40 (0.85) | -0.60 (1.01)
  Week 2 | -0.46 (0.96) | -0.60 (0.90) | -0.72 (1.12) | -1.00 (1.27)
  Week 3 | -0.57 (1.08) | -0.78 (1.02) | -0.84 (1.22) | -1.33 (1.49)
  Week 4 | -0.70 (1.12) | -0.87 (1.13) | -0.94 (1.38) | -1.43 (1.63)
  Week 5 | -0.84 (1.17) | -0.97 (1.20) | -1.06 (1.50) | -1.48 (1.68)
  Week 6 | -0.92 (1.25) | -1.01 (1.32) | -1.13 (1.52) | -1.58 (1.73)
  Week 7 | -1.03 (1.31) | -1.06 (1.40) | -1.13 (1.59) | -1.57 (1.72)
  Week 8 | -1.09 (1.39) | -1.07 (1.49) | -1.26 (1.59) | -1.53 (1.79)
  Week 9 | -1.16 (1.42) | -1.13 (1.49) | -1.27 (1.56) | -1.63 (1.76)
  Week 10 | -1.18 (1.44) | -1.19 (1.56) | -1.33 (1.65) | -1.67 (1.83)
  Week 11 | -1.25 (1.46) | -1.23 (1.57) | -1.36 (1.64) | -1.69 (1.80)
  Week 12 | -1.28 (1.50) | -1.24 (1.60) | -1.36 (1.67) | -1.82 (1.84)
  Week 13 | -1.32 (1.55) | -1.27 (1.63) | -1.43 (1.72) | -1.85 (1.93)
  Week 14 | -1.37 (1.60) | -1.34 (1.74) | -1.47 (1.69) | -1.88 (1.88)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15mg QD; Week 14 change from baseline; Test type: Superiority — DS-5565 20 mg and 30 mg are tested against placebo at significance level of 0.025, respectively. If both arms are statistically significant, DS-5565 15 mg arm will be tested at level of 0.05. If neither of the arms is statistically significant, DS-5565 15 mg arm is no longer tested. If either DS-5565 20 mg or DS-5565 30 mg is statistically significant, DS-5565 15 mg arm is tested at level of 0.025; p = 0.8773, Mixed Models Analysis; Hazard Ratio (HR) = -0.03, 95% CI 2-sided [-0.35 to 0.30]
Statistical Analysis 2: Comparison: Placebo vs DS-5565 20 mg (10 mg BID); Week 14 change from baseline; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3494, Mixed Models Analysis; Hazard Ratio (HR) = -0.15, 95% CI 2-sided [-0.48 to 0.17]
Statistical Analysis 3: Comparison: Placebo vs DS-5565 30 mg (15 mg BID); Week 14 change from baseline; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0027, Mixed Models Analysis; Hazard Ratio (HR) = -0.50, 95% CI 2-sided [-0.82 to -0.17]

2. Secondary Outcome: Change in Visual Analog Scale From Baseline (Week 14) to Week 66 Following Administration of DS-5565 in Participants With Diabetic Peripheral Neuropathic Pain
Description: Visual Analog Scale (VAS) pain is a 10-point assessment tool to measure pain levels, where 0 is defined as 'no pain' and 10 is defined as 'worst possible pain'. Higher VAS pain scores indicate worse outcome.
  In this outcome, the change from baseline in VAS pain is being reported with negative values representing improvements in pain intensity. The larger the negative value (ie. improvement), the greater the improvement in pain intensity.
Time Frame: From baseline (Week 14) to Week 66
Population: Visual analog scale was assessed in all enrolled participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DS-5565 Open-label Extension
Number analyzed (Participants) | 214
units on a scale
  Week 16 | -0.90 (9.190)
  Week 18 | -4.00 (11.140)
  Week 22 | -7.00 (12.690)
  Week 26 | -6.20 (11.430)
  Week 30 | -7.20 (12.620)
  Week 34 | -7.80 (13.260)
  Week 38 | -7.30 (15.230)
  Week 42 | -8.00 (14.420)
  Week 46 | -8.10 (15.780)
  Week 50 | -7.80 (15.100)
  Week 54 | -9.20 (14.360)
  Week 58 | -8.80 (14.940)
  Week 62 | -10.00 (15.390)
  Week 66 | -10.80 (13.950)

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the participant signed the informed consent up to 7 days after the last dose of the study drug (the post-treatment follow-up visit [Visit 11]), up to 2 years 6 months.
Description: A total of 824 participants were included in the Safety Analysis Set. An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory value or abnormal vital sign), symptom, or disease that developed, regardless of relationship to the study drug.
Arm/Group | Placebo | DS-5565 15mg QD | DS-5565 20 mg (10 mg BID) | DS-5565 30 mg (15 mg BID) | DS-5565 Open-label Extension
All-Cause Mortality (participants affected / at risk) | 0/330 | 0/164 | 2/165 | 0/165 | 1/214
Serious Adverse Events (participants affected / at risk) | 11/330 | 4/164 | 8/165 | 11/165 | 24/214
Other Adverse Events (participants affected / at risk) | 101/330 | 60/164 | 62/165 | 84/165 | 141/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=330) | DS-5565 15mg QD (N=164) | DS-5565 20 mg (10 mg BID) (N=165) | DS-5565 30 mg (15 mg BID) (N=165) | DS-5565 Open-label Extension (N=214)
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Perinephric abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Cerebal infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Drowning (General disorders) | 0 | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Peripheral arterial occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=330) | DS-5565 15mg QD (N=164) | DS-5565 20 mg (10 mg BID) (N=165) | DS-5565 30 mg (15 mg BID) (N=165) | DS-5565 Open-label Extension (N=214)
Nasopharyngitis (Infections and infestations) | 42 | 22 | 24 | 27 | 58
Somnolence (Nervous system disorders) | 13 | 14 | 20 | 24 | 20
Dizziness (Nervous system disorders) | 7 | 8 | 14 | 18 | 16
Oedema peripheral (General disorders) | 4 | 8 | 4 | 14 | 24
Weight increased (Investigations) | 2 | 4 | 5 | 11 | 17
Contusion (Injury, poisoning and procedural complications) | 6 | 2 | 3 | 9 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 1 | 3 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 2 | 4 | 1 | 12
Diabetic retinopathy (Eye disorders) | 16 | 7 | 3 | 6 | 25
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 2 | 1 | 18
Constipation (Gastrointestinal disorders) | 8 | 3 | 3 | 5 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4 | 4 | 11
Oedema (General disorders) | 0 | 2 | 1 | 2 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT02318706/Prot_SAP_000.pdf